CLINICAL TRIAL: NCT07030101
Title: A Phase 3 Double-blind, Multicenter, Randomized, Double-blind, Triple-dummy, Controlled Trial to Assess the Efficacy and Safety of a TCA108 in Participants ≥18 Years of Age With Uncontrolled Hypertension
Brief Title: A Study to Investigate Efficacy and Safety of a TCA108 in Participants ≥18 Years With Uncontrolled Hypertension
Acronym: TRÍADE-HA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCA108-III-0124
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bramicar HCT (Active Comparator): The participants must take 1 tablet per day
  Interventions: Drug: Bramicar HCT
- TCA108 (Experimental): The participants must take 1 tablet per day
  Interventions: Drug: TCA108
- Micardis Anlo (Active Comparator): The participants must take 1 tablet per day
  Interventions: Drug: Micardis Anlo

INTERVENTIONS:
Drug: TCA108 — TCA108
  Arms: TCA108
Drug: Bramicar HCT — Bramicar HCT
  Arms: Bramicar HCT
Drug: Micardis Anlo — Micardis Anlo
  Arms: Micardis Anlo

SUMMARY:
The purpose of this study if to evaluate the efficacy and safety of TCA108 in the treatment of hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 years of age or older at the time of signing the informed consent.
2. Participants with a diagnosis of arterial hypertension presenting with SBP ≥ 140 mmHg and ≤ 170 mmHg and DBP ≥ 90 mmHg and ≤ 110 mmHg, confirmed by triplicate measurements from the reference arm at the screening visit.

   d. Participants on dual antihypertensive therapy at a stable dose for at least four weeks prior to screening, meeting the following criterion:

   • Receiving dual therapy with any antihypertensive agents at low or intermediate doses, or a dual combination in which only one of the drugs is at the maximum dose; except for dual therapy involving telmisartan combined with a thiazide diuretic or amlodipine, which will only be allowed when both drugs are at low doses.

   Participants who meet the above criteria at the screening visit must also meet criterion "e" at the randomization visit:
3. Participants with uncontrolled hypertension, confirmed by ambulatory blood pressure monitoring (ABPM) performed during the screening period, defined as SBP ≥ 130 mmHg and DBP ≥ 80 mmHg.
4. Participant is male or female at birth.
5. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   * Not a childbearing potential (CBP) participant as defined below:
   * surgically sterile (documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy as confirmed by review of the participant's medical records, medical examination, or medical history interview), or postmenopausal (defined as no menses for 12 months).
6. If the participant is a female of childbearing potential, they must have a negative urine pregnancy test at the screening visit and the randomization visit and they must be willing to use any of the following highly effective acceptable forms of contraception for the course of the study:

   * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal)
   * progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable)
   * intrauterine device
   * intrauterine hormone-releasing system
   * bilateral tubal occlusion (if not recently performed, should be established, or confirmed if any doubt)
   * vasectomized partner (if not recently performed, should be established, or confirmed if any doubt)
   * complete sexual abstinence (only if this is within the patients preferred lifestyle).
7. Participant is capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

1. Any clinical observation (clinical/physical assessment) or laboratory condition interpreted by the investigator as posing a risk to the participant's involvement in the clinical trial, or the presence of uncontrolled chronic disease(s).
2. Known contraindication or history of hypersensitivity or intolerance to any components of the medications used during the clinical trial.
3. Essential hypertension with DBP > 110 mmHg and/or SBP > 170 mmHg.
4. Participants who have experienced any cardiovascular event (acute myocardial infarction, unstable angina, newly diagnosed stable angina, stroke, unstable congestive heart failure requiring treatment adjustment), undergone revascularization procedure, or vascular surgery within the 6 (six) months prior to screening.
5. Body mass index (BMI) > 45 kg/m².
6. Uncontrolled type 1 or type 2 diabetes mellitus (glycated hemoglobin [HbA1c] > 8.5%).
7. Known heart failure, New York Heart Association (NYHA) Classes III and IV.
8. Coronary artery disease with planned percutaneous intervention within the next 6 months.
9. Current ventricular arrhythmia requiring treatment.
10. Participants with prolonged corrected QT interval (QTc) [male > 450 ms, female > 470 ms] or tachyarrhythmia.
11. Evidence of a secondary form of hypertension, including but not limited to: aortic coarctation, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's disease, pheochromocytoma, polycystic kidney disease.
12. Renal insufficiency with estimated glomerular filtration rate [eGFR] < 30 mL/min (2021 Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] Creatinine Equation), end-stage renal disease requiring dialysis or kidney transplant.
13. Serum potassium levels ≥ 5.5 mEq/L or ≤ 3.5 mEq/L.
14. Alanine aminotransferase (ALT) > 2.5 times the upper limit of normal (ULN), aspartate aminotransferase (AST) ≥ 2.5 × ULN, bilirubin > 2 × ULN.
15. Symptomatic hyperuricemia (history of gout or uric acid stones).
16. Blood dyscrasias.
17. Any chronic inflammatory condition requiring chronic anti-inflammatory therapy.
18. Disease, physical impairment, or mental condition that, in the judgment of the principal investigator, may interfere with study conduct, including outcome assessments.
19. History of malignancy in any organ system, treated or untreated, within the past 5 years, regardless of evidence of local recurrence or metastasis, except for localized basal cell carcinoma of the skin.
20. Any chronic disease that contraindicates participation according to the investigator's judgment.
21. Current treatment with any of the following concomitant medications that may interfere with the evaluation of efficacy, safety, and tolerability:

    * Prolonged treatment (>15 days) with systemic corticosteroids within the 3 months prior to screening. Prolonged systemic corticosteroid use is also prohibited during study participation. Short-term treatment (<5 days) is acceptable during the study.
    * Chronic stable or unstable use of nonsteroidal anti-inflammatory drugs (NSAIDs) other than acetylsalicylic acid, with chronic use defined as ≥1 week of treatment. Intermittent NSAID use is discouraged throughout the study; if necessary, NSAIDs should not be used for more than one week in total. For participants requiring analgesic or antipyretic agents, acetaminophen is recommended during the study.
    * Use of short-acting oral nitrates (e.g., sublingual nitroglycerin) is permitted; however, participants must not take short-acting oral nitrates within 4 hours prior to any study visit/BP assessment and within 4 hours prior to and during ABPM.
    * Use of long-acting oral nitrates (e.g., Isordil) is permitted; however, the dose must be stable for at least 2 weeks prior to screening and maintained throughout the study.
    * Use of sympathomimetic decongestants is permitted; however, not within 1 day prior to any study visit/BP assessment and within 1 day prior to and during ABPM.
    * Use of theophylline is permitted; however, the dose must be stable for at least 4 weeks prior to screening and maintained throughout the study.
    * Use of phosphodiesterase type V inhibitors is permitted; however, participants must abstain from taking these medications within 1 day prior to screening or any subsequent study visit, as well as 1 day prior to and during ABPM.
    * Use of α-blockers is not permitted, except for alfuzosin and tamsulosin for prostatic symptoms, provided the dose is stable for at least 4 weeks prior to screening and maintained throughout the study.
    * Use of drugs acting on the central nervous system (such as antidepressants, antipsychotics, and antiepileptics) is permitted, provided the dose is stable for at least 3 months prior to screening and maintained throughout the study.
22. Research participants who have participated in clinical trial protocols within the past 12 (twelve) months (Resolution CNS 251, August 7, 1997, item III, subitem J), unless the investigator determines that there may be direct benefit to the participant.
23. Participants who do not have an indication for modification of current therapy, in the judgment of the principal investigator or another physician responsible for the participant.
24. Participants who are pregnant, breastfeeding, or planning to become pregnant, or female participants of childbearing potential not using a reliable contraceptive method as described in section 13.2.
25. History of drug or alcohol abuse within the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-11 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline systolic blood pressure (SBP) after 10 weeks of treatment | 10 weeks

SECONDARY OUTCOMES:
Proportion of participants with blood pressure <130/80 mmHg after 10 weeks of treatment | 10 weeks
Proportion of participants with systolic blood pressure (SBP) <130 mmHg or a change from baseline SBP of at least a 10 mmHg decrease after 10 weeks of treatment | 10 weeks
Mean change from baseline diastolic blood pressure (DBP) after 10 weeks of treatment | 10 weeks
Proportion of participants with diastolic blood pressure (DBP) <80 mmHg or a change from baseline DBP of at least a 5 mmHg decrease after 10 weeks of treatment | 10 weeks
Mean change in 24-hour ABPM (Ambulatory Blood Pressure Monitoring) SBP and DBP from baseline after 10 weeks of treatment | 10 weeks
Evaluate the safety of TCA108 in the treatment of hypertension | 12 weeks
  The safety will be evaluated considering the incidence of adverse events (AEs) reported during the study period.

IPD SHARING:
Plan to Share IPD: No